CLINICAL TRIAL: NCT05762510
Title: An Open Label Study Evaluating the Safety and Efficacy of Gene Therapy for Transfusion-dependent β-Thalassemia by Transplantation of Autologous CD34+ Stem Cells Transduced Ex Vivo With a LentiRed Lentiviral Vector (GMCN-508B Drug Product, Also Called LentiRed)
Brief Title: A Study Evaluating the Safety and Efficacy of LentiRed Drug Product in Transfusion-dependent β-Thalassemia [TDT]
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: First Affiliated Hospital of Guangxi Medical University (Other)
Collaborators: Genmedicn Biopharma Ltd. (Unknown)
Responsible Party: Principal Investigator, Yongrong Lai, MD, Director of Hematology Department of First Affiliated Hospital of Guangxi Medical University, First Affiliated Hospital of Guangxi Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-1101-001
Record Dates: First submitted 2022-01-06; First posted 2023-03-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Transfusion Dependent Beta-Thalassemia
Keywords: LentiRed; Beta-Thalassemia; Human Hematopoietic Stem Cell; gene therapy; CD34+
MeSH Terms: conditions — beta-Thalassemia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LentiRed (Experimental): LentiRed Drug Product
  Interventions: Genetic: GMCN-508B (LentiRed)

INTERVENTIONS:
Genetic: GMCN-508B (LentiRed) — LentiRed Drug Product is administered by intravenous infusion following myeloablative conditioning with busulfan.

SUMMARY:
This is a single-arm, open label, single-dose study in subjects with transfusion dependent β-thalassaemia. The study will evaluate the safety and efficacy of autologous CD34+ Human Hematopoietic Stem Cells that was transduced with LentiRed Lentivrial vector.

DETAILED DESCRIPTION:
Subject participation for this study will be 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. The subject himself/herself or one legal guardian/agent of the subject is required to fully understand the study and voluntarily sign a written informed consent.
2. Ages 5 to 35, no gender limitation.
3. The clinical diagnosis of TDT includes β0/β0, β+/β0, βE/β0 and β+/β+ genotypes. TDT was defined as severe anemia in patients with thalassemia (Hb persistent <70 g/L), regular RBC transfusion and standard iron removal therapy to survive for life.
4. Karnofsky Level of Performance (KPS) score ≥70 in adult subjects and Lansky Level of Performance (LPS) score ≥70 in children subjects.
5. Subjects were determined to undergo autologous hematopoietic stem cell transplantation by the principle investigator.
6. Subjects must have been treated and followed for at least the past 2 years in a specialized center that maintained detailed medical records, including transfusion history.

Exclusion Criteria:

1. Hepatitis B virus (HBV) : HbsAg or HbcAb positive, nucleic acid test positive; Hepatitis C virus (HCV) : HCAb positive, nucleic acid test positive; Positive for Human immunodeficiency virus (HIV) antibody or Treponema pallidum (TP) specific antibody; Tuberculosis: positive interferon gamma release test.
2. A white blood cell (WBC) count <3×10^9/L and/or platelet count <100×10^9/L, splenectomy was performed before.
3. Uncured bleeding abnormalities.
4. Any previous or current malignancy, myeloproliferative disease, or immune deficiency disease.
5. Immediate family member with a known or suspected Familial Cancer Syndrome (including but not limited to hereditary breast and ovarian cancer syndromes, hereditary non-polyposis colorectal cancer syndromes and familial adenomatous polyposis).
6. Previous hematopoietic stem cell transplantation (HSCT).
7. Advanced liver disease, defined as: 1) Baseline alanine aminotransferase (ALT) or direct bilirubin ≥3 normal upper limit (ULN), or 2) Liver biopsy demonstrating cirrhosis, any evidence of bridging fibrosis, or acute hepatitis.
8. Baseline estimated glomerular filtration rate (eGFR) < 70 mL/min /1.73 m2, as determined using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) creatinine equation for ≥18 years of age, and Besides Schwartz Equation calculator < 18 years of age.
9. Uncontrolled seizure disorder.
10. Diffusion capacity of Carbon monoxide dispersion (DLco) <50% of predicted (corrected for hemoglobin and or alveolar ventilation, as clinically indicated ).
11. A cardiac T2* <20 ms by magnetic resonance imaging (MRI).
12. Severe iron overload, which in the opinion of the physician is grounds for exclusion.
13. Clinically significant pulmonary hypertension.
14. Participation in another clinical study with an investigational drug within 30 days of screening.
15. Failure to obtain appropriate informed consent.
16. Any other condition that would render the subject ineligible for HSCT, as determined by the attending transplant physician or investigator.
17. Contraindications to the conditioning regimen.
18. Prior receipt of genetic stem cell therapy.
19. Diagnosis of significant psychiatric disorder of the subject that could seriously impede the ability to participate in the study.
20. Pregnancy or breastfeeding in a postpartum female or absence of adequate contraception for fertile subjects. Females of child-bearing potential are required to use effective contraception from the screening period until at least 6 months after drug product infusion. Male subjects are also required to use effective contraception (including condoms) from the screening period until at least 6 months after drug product infusion.
21. Live vaccines were administered within 6 weeks prior to screening.
22. Known history of hypersensitivity to the ingredients used in the trial.
23. An assessment by the investigator that the subject would not comply with the study procedures outlined in the protocol.

Ages: 5 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Estimated)
Dates: Start 2023-02-22 (Actual); Primary Completion 2028-04-01 (Estimated); Study Completion 2030-10-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects who achieved transfusion independence, defined as an average Hb ≥ 9 g/dL without any pRBC transfusions for a continuous period of ≥ 6 months at any time during the study after LentiRed Drug Product infusion. | From time of drug product infusion up to 24 months
  TI was defined as an average hemoglobin (Hb) >= 9 g/dL without any packed red blood cells (pRBC) transfusions for a continuous period of >=6 months at any time during the study after Drug Product infusion.
Number and proportion of subjects who maintained βA-T87Q-globin(HbAT87Q) at ≥2.0 g/dL for ≥ 6 months after LentiRed Drug Product infusion. | From time of drug product infusion up to 24 months
  Percentage of participants with sustained production of >=2.0 grams per deciliter (g/dL) of hemoglobin A (HbA) containing βA-T87Q-globin (HbAT87Q) for 6 months was reported.
Proportion of subjects whose red blood cells (RBC) transfusion requirement was reduced for ≥6 months after LentiRed Drug Product infusion, compared to previous 2-year transfusion records. | From time of drug product infusion up to 24 months
  The annualized number of pRBC transfusions over the 2 year period prior to drug product infusion was compared to the annualized number of pRBC transfusions post drug product infusion and the percentage change was reported.

SECONDARY OUTCOMES:
Proportion of subjects who achieved transfusion independence, defined as an average Hb ≥ 9 g/dL without any pRBC transfusions for a continuous period of ≥ 3 months at any time during the study after LentiRed Drug Product infusion. | From time of drug product infusion up to 24 months
  TI was defined as an average hemoglobin (Hb) >= 9 g/dL without any packed red blood cells (pRBC) transfusions for a continuous period of >=3 months at any time during the study after Drug Product infusion.
Proportion of subjects who achieved Neutrophil engraftment. | From time of drug product infusion up to 24 months
  Neutrophil engraftment was defined as achieving 3 consecutive absolute neutrophil count (ANC) >= 0.5 × 10^9/L on different days after a post-transplant value of < 0.5 × 10^9/L within 42 days after drug product infusion.
Incidence of transplant-related mortality through 100 days post drug product infusion. | Through 100 days post-Drug Product infusion
  Transplant-related mortality was determined by the investigator (any deaths considered related to the transplant.)
Overall survival. | From time of drug product infusion up to 24 months
  Overall survival was defined as time from date of LentiRed Drug Product infusion (Day 0) to date of death.
Detection of vector-derived replication competent lentivirus (RCL) in any subject. | From time of drug product infusion up to 24 months
  Blood samples were analyzed for detection of RCL
Characterization of events of insertional mutagenesis leading to clonal dominance or leukemia. | From time of drug product infusion up to 24 months
  Linear amplification-mediated polymerase chain reaction (LAM-PCR) coupled with next generation sequencing and subsequent (semi-) automated data mining allowed high-throughput analysis of vector integration site (IS) in blood cells from treated participants at multiple time points. ISs detected in peripheral blood cells at early time points generally were due to the expansion of transduced short-term progenitor stem cell clones, and gradually shift to include sites detected due to expansion of transduced long-term stem cell clones. An efficient transduction procedure was anticipated to give rise to a polyclonal population in the participant, reflected by the detection of multiple IS. Additionally, ISA allowed monitoring of the relative contribution of individual clones over time. Number of participants who had IS that contributed to >=30% of the total clones at any time was used as a first step to investigating whether clonal dominance was achieved.
Monitor of frequency of clinical adverse events (AEs). | From signing of informed consent to 24 months after the drug product infusion
  An AE was defined as any unfavorable and unintended sign (including abnormal laboratory findings), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Therapeutic globin expression, as measured by assessing the ratio of βA-T87Q-globin to α -globin in whole blood, as well as the amount of βA-T87Q-globin to as a fraction of all β -chains in whole blood. | From time of drug product infusion up to 24 months
  globin expression measured by HPLC
Average vector copy number (VCN) in cell populations from peripheral blood and bone marrow containing the integrated LentiRed lentiviral vector. | From time of drug product infusion up to 24 months
  VCN will be monitored after drug product transfusion

CONTACTS AND LOCATIONS:
Locations (1):
- The affiliated hospital of guangxi medical university, Nanning, Guangxi, China

IPD SHARING:
Plan to Share IPD: No